CLINICAL TRIAL: NCT03900364
Title: Robot-assisted Partial Nephrectomy Versus Laparoscopic Partial Nephrectomy: A Prospective, Randomised, Single-blind Trial Comparing Two Surgical Techniques
Brief Title: a Prospective Trial Comparing Robot-assisted Partial Nephrectomy Versus Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Lukas Oberhammer, Principal Investigator, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT2019
Record Dates: First submitted 2019-02-12; First posted 2019-04-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Renal Cell; Renal Malignant Tumor; Renal Cyst; Renal Tumor
Keywords: partial nephrectomy; robot-assisted partial nephrectomy; laparoscopic partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted partial nephrectomy (Other): partial nephrectomy performed with the da Vinci Surgical System
  Interventions: Procedure: partial nephrectomy
- laparoscopic partial nephrectomy (Other): partial nephrectomy performed with conventional laparoscopic surgery
  Interventions: Procedure: partial nephrectomy

INTERVENTIONS:
Procedure: partial nephrectomy — Partial nephrectomy is the standard technique for organ-sparing resection of renal tumors. The EAU Guidelines recommend partial nephrectomy to all patients with T1 tumours and can be performed either with an open, pure laparoscopic or robot-assisted approach, based on surgeon's expertise and skills.

SUMMARY:
In this trial the investigators want to examine and compare oncological and surgical outcomes of two surgical techniques in a prospective, randomised, single-blind trial. Therefore the investigators are going to include 30 patients with a renal mass who need surgical treatment. When they fulfill the inclusion criteria they get randomised either for robot-assisted partial nephrectomy or laparoscopic partial nephrectomy. Primary endpoint is the oncological outcome (residual tumor classification, TNM classification), secondary endpoints are operation time, time of ischemia, blood loss, pain after surgery, kidney function, complications and hospital stay.

DETAILED DESCRIPTION:
All patients taking part in the study are first given a R.E.N.A.L. nephrometry score. Based on that score they are allocate to either of :

cohort I (low complexity of the tumour) or cohort II (intermediate complexity of the tumour).

Thereafter, the patient will be randomly placed into either to laparoscopic partial nephrectomy or robotic-assisted partial nephrectomy. Both these surgical techniques are well established and standardized procedures to remove a renal mass.

Preoperatively, the preparation is nearly the same for both techniques. The patient is positioned in flank position with the affected side up.

Thereafter:

Pneumoperitoneum is achieved with a Veress needle and trocars which are placed under direct vision. The only difference between the two techniques is the number of trocars, performing the laparoscopic partial nephrectomy three or four ports are used, performing the robotic-assisted partial nephrectomy five ports are used.

Intraabdominal, the kidney is exposed by incising along the Toldt line to moblize the colon. After exposing the ureter and the gonadal vein dissection is continued proximally toward the renal hilum. Following this, Gerota's fascia is incised to expose the tumour and the surrounding renal capsule. Now the renal artery has to be clamped to avoid bleeding followed by excision of the tumour. The surgery takes about three hours, the complication rate is more the same for both techniques.

Primary endpoint is the resection margin to see if there are any difference between the two surgical techniques.

Information about the resection margin and pathological staging will be given through our pathological department. The histological examination normally takes about five to seven days.

Further parameters are taken by following schema:

Information about age, sex, body mass index, other diseases and medication is documented on the day of inpatient admission.

Blood samples for haemoglobin and kidney function are taken at the day of inpatient admission, four hours after surgery, first day after surgery and the day of discharge from hospital.

The duration of surgery is documented throughout the operative protocol. R.E.N.A.L Nephrometry score is evaluated preoperative, to be able to compare the complexity of surgery.

Renal ischemia is documented throughout the operative protocol. Blood loss is documented during surgery. Pain is documented with the aid of the visual analogue scale (VAS Scale). This will be evaluated four hours after surgery, day one after surgery, day two after surgery and on the day of discharge from hospital.

Complications are documented with the aid of the clavien-dindo classification. Three follow-ups will be performed. The first follow-up will be held two weeks after surgery to discuss the histological result and examine haemoglobin, kidney function and pain. The second follow-up will be held six months after surgery, the third follow-up 12 months after surgery. At this time a re-examination again haemoglobin and kidney function will be performed as well as a computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years
* solid renal mass suspicious for renal cell carcinoma or at least Bosniak III cyst
* signed informed consent

Exclusion Criteria:

* performed kidney surgery at the same side
* Pregnancy
* RENAL Nephrometry score III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with R0 status | one year
  The tumor status following further treatment is described by the residual tumor classification. R0 means no residual tumor, R1 means microscopic residual tumor. The investigators are going to examine if there are any significant differences concerning tumor status between these two surgical techniques

SECONDARY OUTCOMES:
Operation time | one year
  time of surgery (in minutes)
Ischemia time | one year
  Time of warm ischemia during laparoscopic or robot-assisted partial nephrectomy
Blood loss | one year
  The amount of blood loss during performing partial nephrectomy
Postoperative pain | one year
  Postoperative pain is going to be documented with the aid of the visual analogue scale. The visual analogue scale is a validated, subjective measure for pain. With the aid of a scale from zero to ten which represents a continuum between 'no pain' (0) and 'worst pain' (10) the subjective pain of each participant will be evaluated. This will be done four hours after surgery, day one after surgery, day two after surgery and on the day of discharge from hospital.
Kidney function | one year
  Before and after surgery blood samples are taken to evaluate the kidney function with the aid of Serum creatinine and the glomerular Filtration rate
Complications | one year
  Postoperative complications evaluated by 'clavien-dindo' classification
Hospital stay | one year
  The length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinikum Salzburg, Department for Urology and Andrology, Salzburg, Austria